CLINICAL TRIAL: NCT03132116
Title: Intra-nodal Injection of Gentamicin for the Treatment of Suppurated Cat Scratch Disease's Lymphadenitis: A Randomized Controlled Study
Brief Title: Intra-nodal Injection of Gentamicin for the Treatment of Suppurated Cat Scratch Disease's Lymphadenitis
Acronym: BIGG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15 7834 08
Record Dates: First submitted 2017-03-05; First posted 2017-04-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Cat-Scratch Disease
Keywords: Cat Scratch Disease's lymphadenitis; Infectious Diseases
MeSH Terms: conditions — Cat-Scratch Disease; Communicable Diseases | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentamicin (Experimental): intra-nodal injection of gentamicin
  Interventions: Drug: gentamicin
- Placebo (Placebo Comparator): intra-nodal injection of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: gentamicin — After inclusion in the study, patient will be randomized. According to randomization, patient will receive an intra-nodal injection of gentamicin .
  As well, azithromycin will be prescribed for all patients for 5 days. Patients will be followed-up each week until week 4 (Day 28).
  Arms: Gentamicin
Drug: placebo — After inclusion in the study, patient will be randomized. According to randomization, patient will receive an intra-nodal injection of placebo.
  As well, azithromycin will be prescribed for all patients for 5 days. Patients will be followed-up each week until week 4 (Day 28).
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
To compare effect of intra-nodal injection of gentamicin versus placebo on the outcome at 28 days of suppurated cat scratch disease's (CSD) lymphadenitis treated by oral azithromycin.

DETAILED DESCRIPTION:
Double blind controlled study versus placebo. Patients with suppurated CSD's lymphadenitis will receive immediately after the pus aspiration (performed for a diagnostic purpose) an intra-nodal injection of gentamicin or of placebo (NaCl 0,9%) and be treated with oral azithromycin for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Suppurated CSD's adenitis:

  * Suppurated form of adenitis confirmed by echography
  * Serology positive for Immunoglobulin G and/or Immunoglobulin M against B. henselae

Exclusion Criteria:

* Suppurated adenitis non related to CSD
* Non-suppurated CSD's adenitis
* Suppurated CSD's adenitis already fistulized
* Suspected visceral B. henselae infection (neurologic or ophthalmic symptoms, hepato-splenic or valvular involvement confirmed by echography)
* Immunodepression (except diabetes)
* Pregnancy
* Contraindication to pus aspiration from lymphadenitis (history of bleeding or patient taking curative anticoagulation therapy or platelet count < 50.000/mm3)
* Contraindication to azithromycin (history of QT interval prolongation, history of liver toxicity of hypersensitivity to macrolides or treatment with ergotamine, dihydroergotamine, bepridil, cisapride, pimozide, mizolastine or colchicine) or to aminoglycosides (myasthenia, history of hypersensitivity to aminoglycosides).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency at day 28 of CSD's adenitis favorable outcome | Day 28
  Adenitis favorable outcome characterized as : Reduction of the volume of the adenitis, Without requirement of supplementary needle aspirations after day 7's visit, And without requirement of a surgical excision or incision of the adenitis.

SECONDARY OUTCOMES:
Reduction of the adenitis | from Day 0 to Day 28
  Percentage of volume reduction of the adenitis
Evaluation of the pain related to the adenitis | between Day 0, Day 7 and Day 28
  Percentage of reduction of the pain related to the adenitis
Fistulization of the adenitis | Day 7 and day 28
  Number of patients with persisting cutaneous fistulization of the adenitis
Surgical action | Day 28
  Number of patients requiring surgical excision or incision of the adenitis
Protein C reactive | Day 0 and day 7
  Percentage of decrease of serum Protein C reactive
Antibiotic resistance | Day 28
  Genotypic profile of resistance to macrolides and aminoglycosides
Safety of treatment | Day 7 and day 28
  Incidence of Treatment-Emergent Events linked to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MARTIN-BLONDEL, MD, PhD, Principal Investigator — University Hospital of Toulouse, Infectious & Tropical Diseases department
Locations (21):
- France (21):
  - Albi Hospital, Albi
  - Amiens-Picardie Hospital, Amiens
  - Angers Hospital, Angers
  - Auch Hospital, Auch
  - Bordeaux University Hospital, Bordeaux
  - Cahors Hospital, Cahors
  - Castres Hospital, Castres
  - Vendée Hospital, La Roche-sur-Yon
  - Limoges University Hospital, Limoges
  - Hospices Civils Lyon, Lyon
  - Montauban Hospital, Montauban
  - Montpellier University Hospital, Montpellier
  - Nîmes University Hospital, Nîmes
  - Pau Hospital, Pau
  - Perpignan Hospital, Perpignan
  - Rennes Hospital, Rennes
  - Rodez Hospital, Rodez
  - Saint-Brieuc Hospital, Saint-Brieuc
  - Saint-Nazaire Hospital, Saint-Nazaire
  - Tarbes Hospital, Tarbes
  - Microbiology Laboratory, Toulouse

IPD SHARING:
Plan to Share IPD: No